CLINICAL TRIAL: NCT03043378
Title: Chronic Non-Malignant Pain in Cancer Patients at a Supportive Care Clinic
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0901; NCI-2018-01268 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Malignant Neoplasms of Independent (Primary) Multiple Sites; Non-malignant pain; Supportive care; Questionnaires; Surveys; Chronic non-malignant pain
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Non-Malignant Pain - Cancer Patients: Chronic non-malignant pain among cancer patients undergoing a consultation at the outpatient Supportive Care Clinic at MD Anderson Cancer Center.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete three questionnaires at consultation visit.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn how frequently cancer patients in the Supportive Care Center have chronic, non-malignant pain. Chronic, non-malignant pain is pain that is neither related to cancer nor its treatment and lasts beyond the normal tissue healing time of 3 months.

DETAILED DESCRIPTION:
If participant is found to be eligible and agrees to take part in this study, participant will be asked to complete 3 questionnaires about participant's pain, pain level, and what drugs participant takes to treat participant's pain. Participant will also be asked a few questions about tobacco use. These questionnaires should take about 20 minutes to complete.

Researchers will also collect information from participant's medical record such as participant's date of birth, sex, race, marital status, economic background, and medical history.

Length of Study:

Participation on this study will be over after participant has completed the last questionnaire.

This is an investigational study.

Up to 200 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer with or without active disease
2. Consultation visit at an outpatient supportive care clinic
3. Age 18 or greater
4. Report of having pain within the last 3 months

Exclusion Criteria:

1) Memorial Delirium Assessment Scale >13

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing consultation at the Supportive Care Clinic at MD Anderson Cancer Center.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Frequency of Chronic Non-Malignant Pain Among Cancer Patients | 1 day
  Frequency assessed by Edmonton Symptom Assessment Scale (ESAS-FS)
Frequency of Chronic Non-Malignant Pain Among Cancer Patients | 1 day
  Frequency assessed by Brief Pain Inventory.
Frequency of Chronic Non-Malignant Pain Among Cancer Patients | 1 day
  Frequency assessed by the Charlson Comorbidity Index.
Frequency of Chronic Non-Malignant Pain Among Cancer Patients | 1 days
  Frequency assessed by Pain Characteristic Survey.
Frequency of Chronic Non-Malignant Pain Among Cancer Patients | 1 day
  Frequency assessed by Karnofsky Performance Scale.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org